CLINICAL TRIAL: NCT05563350
Title: Association Between Variations in CYP Pheno- and Genotypes and Plasma Concentration of Chlordiazepoxide in the Treatment of Alcohol Withdrawal Symptoms
Brief Title: Metabolism of Chlordiazepoxide in the Treatment of Alcohol Withdrawal Symptoms
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Nanna Reiter, Principal investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: KLOPOXID2021
Record Dates: First submitted 2022-09-01; First posted 2022-10-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2022-09

CONDITIONS: Alcohol Withdrawal
Keywords: ICU; Intensive care; CYP3A4; CYP2C19; Chlordiazepoxide
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Blood samples — p-chlordiazepoxide and metabolites, p-omeprazole and metabolites, p-midazolam and metabolites, CYP3A4 and CYP2C19 genotyping
  Other Names: Midazolam and omeprazole as pharmacological probes

SUMMARY:
The aim of this study is to elucidate if CYP-phenotypes, variations in CYP-genotypes and dose of chlordiazepoxide is correlated to chlordiazepoxide plasma concentrations in patients admitted to Intensive Care or High Dependency Units due to either respiratory insufficiency and/or agitation while treated for alcohol withdrawal symptoms.

DETAILED DESCRIPTION:
Pharmacological treatment caries a risk of overdosing and adverse events. Chlordiazepoxide, among other sedative drugs, has been associated with an increased risk of death. Chlordiazepoxide treatment for alcohol withdrawal symptoms will render some patients in need of ventilatory support and ICU admission. Other patients will not obtain the desired effect from the treatment and will be in a state of agitation despite having received high doses of chlordiazepoxide. This individual variation in effect is not predictable and may be explained by variations in the capacity of drug metabolism.

Chlordiazepoxide is extensively metabolized in the liver by hepatic microsomal enzymes and exhibits capacity limited, protein binding sensitive, hepatic clearance. Metabolism is primarily by cytochrome P450 (CYP), especially CYP3A4 and CYP2C19 systems. Evaluation of CYP phenotypes by drug probe phenotyping is extensively used. Midazolam possesses several characteristics that makes it useable as a pharmacological probe for CYP3A activity despite having already received other benzodiazepines. It is metabolized to a primary metabolite exclusively by CYP3A4/3A5.Omeprazole can likewise be used as a pharmacological probe for CYP2C19.

The drug of investigation is chlordiazepoxide, which has been given before study inclusion. After inclusion and during the study period (12 hours), it is not allowed to administer chlordiazepoxide to the patient. In case of abstinence, the recommended therapy is diazepam or propofol.

Blood samples will be collected and plasma concentrations of chlordiazepoxide and metabolites will be analyzed and compared with the amount of chlordiazepoxide administered at inclusion and 12 hours after inclusion.

Independent variables:

* Variations in genotypes of CYP3A4/3A5 and CYP2C19.
* Phenotypes of CYP3A4/3A5 and CYP2C19, analyzed as above /below the median value of enzyme activity.

Variations in genotypes of CYP3A4/3A5 and CYP2C19 will be analyzed from blood samples.

Phenotyping of CYP3A4/3A5 and CYP2C19 will be performed with midazolam and omeprazole as pharmacological probes respectively. 2 mg of midazolam and 10 mg of omeprazole will be administered intravenously as bolus within 12 hours after inclusion. Blood samples 2 h after dosing (t=2 h dosing) will be collected and analyzed for plasma concentrations of omeprazole, hydroxyomeprazole, midazolam and 1-hydroxymidazolam. The ratio between omeprazole and hydroxyomeprazole will be used to classify the CYP2C19 phenotype as the ratio between midazolam and 1-hydroxymidazolam will be used in the classification of CYP3A4/3A5

By measuring concentration of chlordiazepoxide and the ability to metabolize chlordiazepoxide in ICU- or HDU-patients with respiratory insufficiency, impaired consciousness or agitation after treatment for alcohol withdrawal symptoms, we will investigate if there is a correlation between the patient's phenotypes of the CYP3A4/3A5 and CYP2C19 systems (independent variable) and the concentration of chlordiazepoxide (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Treatment with minimum 200 mg chlordiazepoxide for alcohol withdrawal symptoms during hospital admission
* Acute admittance to ICU or HDU due to respiratory insufficiency, impaired consciousness or agitation.
* Inclusion possible within 12 h of ICU/HDU admission.

Exclusion Criteria:

* Allergies to omeprazole/esomeprazole and midazolam
* Treatment with chlordiazepoxide within the first 12 h after inclusion (from blood samples at inclusion until blood samples 12 h after inclusion)
* Treatment with omeprazole/esomeprazole within 1 day prior to ICU/HDU admission and within the first 12 h after inclusion.
* Treatment with midazolam within 1 day prior to ICU/HDU admission
* Cardiac arrest prior to admission
* Pregnancy (a negative hcg (from urine or blood sample) has to be present before inclusion of women aged <50 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 26 consecutive patients will be included no later than 12 h after ICU or HDU admission after treatment with moderate or large doses (minimum dose 200 mg independently of body weight) of chlordiazepoxide for alcohol withdrawal symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-01-29 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of chlordiazepoxide and metabolites | At inclusion and 12 hours after inclusion
  p-chlordiazepoxide and metabolites.

SECONDARY OUTCOMES:
Half-life (T½) for chlordiazepoxide | At inclusion and 12 hours after inclusion
  Half-life (T½) for chlordiazepoxide will be estimated from the area under the concentration time curve (AUC) from concentrations of chlordiazepoxide at inclusion and 12 hours after inclusion.
Cumulative dose of chlordiazepoxide before admission to ICU/HDU | From date of hospital admittance until the date of inclusion in the study no later than 12 hours after admission on either ICU or HDU
  Chlordiazepoxide dose in mg
ICU/HDU and hospital length of stay (LOS) within 90 days | 90 days after ICU admission and 90 days after hospital admission
  ICU Length of stay and Hospital length of stay
Need for mechanical ventilation within 90 days | 90 days after inclusion
  Duration of treatment with mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Reiter, MD, Principal Investigator — Bispebjerg and Frederiksberg Hospital
Locations (1):
- Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided